CLINICAL TRIAL: NCT02686619
Title: Multicentre, Prospective, Randomized, Open-label Study Comparing the Efficacy and Safety of CellCept With Delayed Introduction of Sirolimus and Discontinuation of Cyclosporine, With Those of Standard Immunosuppression Comprising CellCept and Long-term Continuation of Cyclosporine in Renal Transplant Recipients Receiving Induction by Zenapax and Treated With Corticosteroids for 8 Months
Brief Title: Study Comparing Efficacy and Safety of Mycophenolate Mofetil (Cellcept) With Delayed Introduction of Sirolimus and Discontinuation of Cyclosporine, With Those of Mycophenolate Mofetil and Long Term Continuation of Cyclosporine in Renal Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18326
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Cyclosporine; Daclizumab; Mycophenolic Acid; Prednisolone; Sirolimus

ARMS (2):
- Mycophenolate Mofetil + Cyclosporine (Active Comparator): Participants will receive mycophenoate mofetil, daclizumab, cyclosporine, and corticosteroids (prednisolone) for 3 to 12 months.
  Interventions: Drug: Cyclosporine; Drug: Daclizumab; Drug: Mycophenoate Mofetil; Drug: Prednisolone
- Mycophenolate Mofetil + Sirolimus (Experimental): Participants will receive mycophenoate mofetil, daclizumab, and corticosteroids (prednisolone) for 3 to 12 months. Participants will also receive cyclosporine which will be replaced with sirolimus at later stage of the study.
  Interventions: Drug: Cyclosporine; Drug: Daclizumab; Drug: Mycophenoate Mofetil; Drug: Prednisolone; Drug: Sirolimus

INTERVENTIONS:
Drug: Cyclosporine — Cyclosporine tablets orally once daily at dose level adapted to maintain concentration at 2 hours after administration (C2): 1000-1500 nanogram per milliliter (ng/mL) during Day 0 to Week 4, and 800-1200 ng/mL during Week 4 to Week 52. For Mycophenoate Mofetil + Sirolimus treatment arm, at Week 12, dose of cyclosporine will be reduced by 50% for 3 days, followed by 1/4 of the dose for 3 days, and then cyclosporine will be stopped.
  Other Names: Neoral
Drug: Daclizumab — Daclizumab 2 milligram (mg) per kilogram (kg) will be administered as intravenous infusion over 15 minute on Day 0 (during the 24 hours preceding renal transplantation) and at a dose of 1 mg/kg on Day14.
  Other Names: Zenapax
Drug: Mycophenoate Mofetil — Mycophenoate mofetil 1 gram (g) (2*500mg tablets or 4*250mg capsules) will be given twice daily (daily dose of 2 g) orally for 12 months.
  Other Names: CellCept
Drug: Prednisolone — Prednisolone 250 mg intravenously on Day 0, followed by 0.5 mg/kg orally daily (maximum 40 mg daily) from Day 1 to Day 7, then 0.25 mg/kg orally daily (maximum 20 mg daily), then dose will be stepwise reduced by 2.5 mg per week to reach to a dose level of 10 mg daily and continued up to 6 months and finally drug will be discontinued after 8 months.
  Other Names: Solupred
Drug: Sirolimus — Sirolimus tablets will be given orally from week 12 to week 52, starting with loading dose of 10 mg daily for 2 days followed by 6 mg daily to adapt to trough concentrations of 8-15 ng/mL from week 12 to week 39, and 5-10 ng/mL from week 39 to week 52.
  Other Names: Rapamycin
  Arms: Mycophenolate Mofetil + Sirolimus

SUMMARY:
This multicentre, prospective, randomized, open-label study will compare the safety and efficacy of mycophenolate mofetil with delayed introduction of sirolimus and discontinuation of cyclosporine, with those of mycophenolate mofetil and long term continuation of cyclosporine in renal transplant recipients receiving daclizumab (Zenapax) as induction treatment and followed by 8 month treatment with corticosteroids. The anticipated time on study treatment is 12 months. Participants who will complete the initial 12-month study and who will provide written informed consent will be eligible to participate in a 60-month follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of a first cadaveric kidney graft
* Antilymphocyte antibodies and panel reactive antibodies (PRA) less than 30 percent (%) (historical peak and/or current value)
* Cold ischaemia time less than or equal to 36 hours

Exclusion Criteria:

* Kidney from a living donor; donor greater than (>) 65 years of age; second renal graft, or more; or multiple organ transplant
* Known hypersensitivity to any of the drugs in the study or their components
* History of cancer or malignancy during previous 5 years, other than successfully treated spinocellular or basal cell cancer
* Participant presenting, on inclusion, either symptoms suggestive of active gastroduodenal ulcer, or gastroduodenal ulcer confirmed by fibroscopy and biopsy, and requiring treatment
* Participant with severe refractory hyperlipidaemia
* Pregnant woman or nursing mother

Exclusion Criteria for Follow-up Phase:

* Episode of acute rejection greater than or equal to grade I (Banff classification)
* Estimated creatinine clearance (CrCl) at week 12 less than (<) 40 milliliter per minute (mL/min) (Cockcroft-Gault formula)
* Serum creatinine variations >30% during the 15 days before randomization
* Proteinuria >1 gram/24 hour, or mean mycophenolate mofetil dose < 1.5 gram/day during the week before randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2004-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Creatinine Clearance Calculated and Corrected According to Cockcroft Gault at Month 60 | 60 months
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 12 months
Number of Participants With Serious Adverse Events (SAEs) | From 12 months up to 60 months
Creatinine Clearance Calculated and Corrected According to Cockcroft Gault at Week 52 | 52 weeks
Number of Participants With Cancers and Lymphoproliferative Syndromes | Up to approximately 12 months
Number of Participants With Premature Discontinuations due to Adverse Events (AEs) | Up to approximately 12 months
Change From Baseline in 24-Hour Urinary Protein at Week 52 | 52 weeks

SECONDARY OUTCOMES:
Mean Inverse Creatinine Concentration | Week 4, 8, 12, 14, 16, 26, 39, and 52
Creatinine Clearance Calculated and Corrected According to Cockcroft-Gault | Week 4, 8, 12, 14, 16, 26, 39, and 52
Glomerular Filtration Rate (GFR) Measured by Iohexol Clearance | Baseline, Week 52
Number of Participants with Response to Treatment, Defined as Creatinine Clearance >/=60 mL/min at Week 52 | Week 52
Number of Participants With Treated Rejections | Baseline up to Week 52
Mean Serum Creatinine Concentration | Week 4, 8, 12, 14, 16, 26, 39, and 52
Number of Participants With Biopsy-proven Acute Rejections | Baseline up to Month 60
Number of Participants With Histologic Evaluation of the Graft | Week 52
Number of Participants Who Were Alive | Month 60
Number of Participants With Graft Survival | Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (15):
- France (15):
  - Angers
  - Caen
  - Clermont-Ferrand
  - La Tronche
  - Lille
  - Limoges
  - Lyon
  - Paris
  - Poitiers
  - Reims
  - Rennes
  - Rouen
  - Salouël
  - Strasbourg
  - Tours